CLINICAL TRIAL: NCT07115251
Title: Plans4Care: Personalized Dementia Care on Demand
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Plans4Care Inc (Industry)
Collaborators: Drexel University (Other); Thomas Jefferson University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sokha Koeuth, MPI, Plans4Care Inc
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2306009970; 4R44AG084365 (NIH)
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Dementia; Dementia Alzheimer Type; Alzheimer Dementia (AD); Memory Loss
Keywords: Caregiver, Dementia, Memory Loss, Alzheimer
MeSH Terms: conditions — Dementia; Alzheimer Disease; Memory Disorders

STUDY DESIGN:
Intervention Model Description: This is a non-drug intervention that provides caregivers of people with dementia education and actionable non-drug strategies. Caregivers also have access to speak with a care advisor for additional tele-support.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- initial treatment group (Experimental): Receives Plans4Care web app
  Interventions: Behavioral: Plans4Care
- Waitlist control (Other): At 6 months, receives access to the Plans4Care web app
  Interventions: Behavioral: Plans4Care

INTERVENTIONS:
Behavioral: Plans4Care — Caregivers assigned to treatment condition will receive: 1) access to the web-app; 2) an orientation to the web-app involving initial set up; and 3) a brief video explaining use of the web-app. Caregivers will be guided through accessing the platform, creating an account and completing a brief set of background questions.
  Other Names: P4C

SUMMARY:
The Plans4Care study is a research study funded by the National Institute on Aging (Grant# R44AG084365). The Plans4Care app is designed to help family caregivers address over 90 common care challenges such as behavioral symptoms (anxiety, agitation), functional changes and other concerns, and receive an action plan which provides easy-to-use non-drug strategies, resources, tips and education.

The goal of the study is to evaluate whether using the Plans4Care app will help you feel more confident providing care to your family member with dementia, better understand dementia, and enhance your own well-being. You also have the option to talk with a care advisor who can practice use of strategies or address concerns you may have.

DETAILED DESCRIPTION:
We invite caregivers of people with dementia to take part in this research study. You are being asked to evaluate a new online application (web app) called Plans4Care that provides personalized action plans to address common dementia-related care challenges including tips for your own health and wellbeing. This study is being conducted by Plans4Care, Inc. and researchers at Drexel University in collaboration with Thomas Jefferson University.

Participants who are eligible for this study are:

1. A family, friend, or neighbor who self-identifies as having primary care responsibilities for a person with memory loss;
2. >21 years of age;
3. Able to use an internet capable device (computer, tablet or smart phone), and have stable internet access;

6. Actively (e.g., past 6 months) managing a dementia-related care challenge.

ELIGIBILITY:
Inclusion Criteria:

1. A family, friend, or neighbor who self-identifies as having primary care responsibilities for a person with memory loss;
2. >21 years of age;
3. Able to use an internet capable device (computer, tablet or smart phone), and have stable internet access;

6. Actively (e.g., past 6 months) managing a dementia-related care challenge.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Caregiver well-being | Baseline, 3 months, 6 months and 12 months
  13-item validated Perceived Change for Better Index assesses caregiver perceived change (gotten worse-a little/a lot, stayed the same, improved-a little/a lot) in affect, somatic, manage daily care.

SECONDARY OUTCOMES:
Caregiver/customer satisfaction (outcome) Net promoter Score | 6 months and 12 months
  "How likely is it that you would recommend Plans4Care to a friend or colleague?" (0=not at all to 10=extremely likely). Promoters = score 9 or 10; Passives = score 7 or 8. Detractors = score=0 to 6
Caregiver satisfaction survey | 6 months and 12 months
  A questionnaire designed to gauge how satisfied caregivers are with their work, including their work environment, support systems, and overall job satisfaction.
Health care utilization | Baseline, 3 months, 12 months
  Caregiver report 911 calls, emergency room visits, hospitalizations, nursing home placement for person with AD/ADRD
  Electronic records from primary care practices of emergency room visits and days hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Sokha Koeuth, DHSc, Principal Investigator — Plans4Care Inc; Eric Jutkowitz, PhD, Principal Investigator — Plans4Care Inc; Laura N. Gitlin, PhD, FGSA,FAAN, Study Director — Drexel University; Catherine V Piersol, PhD, OTR/L,FAOTA, FNAP, Study Director — Thomas Jefferson University

IPD SHARING:
Plan to Share IPD: Undecided